CLINICAL TRIAL: NCT02109588
Title: Early Prevention of Childhood Obesity: an Active Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, María Perales Santaella, PhD student, Technical University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prevention childhood obesity
Record Dates: First submitted 2014-03-31; First posted 2014-04-10 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2013-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Sedentary pregnant women
- Exercise group (Experimental): Supervised physical conditioning program of three 55-60 minute sessions per week during whole pregnancy (from week 9 to 38). Each session consists of 25-30 minutes of cardiovascular exercise,10 minutes of specific exercises (strength and balance exercises), and 10 minutes of pelvic floor muscles training
  Aerobic activity was prescribed at light to moderate intensity, aiming for 55-60% of heart rate reserve. All subjects wore a heart rate (HR) monitor (Polar FT7) during the training sessions to ensure that exercise intensity was light to moderate
  Interventions: Behavioral: A supervised physical exercise program

INTERVENTIONS:
Behavioral: A supervised physical exercise program — Supervised physical conditioning program of three 55-60 minute sessions per week during whole pregnancy (from week 9 to 38). Each session consists of 25-30 minutes of cardiovascular exercise,10 minutes of specific exercises (strength and balance exercises), and 10 minutes of pelvic floor muscles training
  Aerobic activity was prescribed at light to moderate intensity, aiming for 55-60% of heart rate reserve. All subjects wore a heart rate (HR) monitor (Polar FT7) during the training sessions to ensure that exercise intensity was light to moderate
  Arms: Exercise group

SUMMARY:
The main aim of this study was to examine the effect of a supervised physical exercise program on the prevention of childhood obesity and its impact on the motor development of the offspring.

DETAILED DESCRIPTION:
The environment where the fetus growths up is essential for the risk of developing some diseases in later life, such as obesity. Exercise has showed being useful in the prevention on excessive maternal weight gain which is linked to fetus weight.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines
* Being able to communicate in spanish
* Giving birth at Hospital Universitario de Torrejón, hospital Universitario de Puerta de Hierro and Hospital Universitario Severo Ochoa (Madrid).

Exclusion Criteria:

* Multiparity
* Obstetrician complications
* Being interested in the study after 16 weeks
* Not being regular in physical exercise program
* Younger than 18 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1100 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Body mass index of the offsprings | 0-24 postpartum months
  Body mass index was measured several times from 0 to 24 months
Fetus body composition | 0-24 postpartum months
  Fetus body composition (percentage of fat) was measured several times from 0 to 24 months
Change from baseline in Maternal gestational weight gain | 40-42 weeks of gestation
  Maternal weight gain during pregnancy
Changes in Baby motor development | 0-24 postpartum months
  Baby motor development was measured after delivery
Recovery time to pre-gestational weight | 6-12 postpartum months
  The time needed to recovery the pre-gestational weight was assessed.
Glycemia level of the offsprings | 0-24 postpartum months
  Glycemia level of the offsprings was measured until 24 months
Postpartum depression | 0-12 postpartum months
  The level of maternal depression was measured after delivery
Change from baseline in Body image satisfaction | up to 36 weeks
  Body image satisfaction was measured during and after pregnancy
Changes from baseline in maternal quality of life | up to 36 weeks
  Maternal quality of life was measured during and after pregnancy
Placenta measurements | At delivery
  Placenta measurements were collected at labor

SECONDARY OUTCOMES:
Maternal outcomes | At delivery
  Type of labor, stage of labor and some other maternal variables were measured at delivery
Control of physical activity | up to 10 weeks
  Control the level of physical activity during and after pregnancy
Changes from delivery in Health of the offspring | 0-24 postpartum months
  Health of the baby included the measurement of other variables such as blood pressure and cholesterol of the offsprings until 24 months
Fetus outcomes | At delivery
  Fetus outcomes were measured at delivery: Apgar score, PH umbilical cord, size and height of the baby, head circumference

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Barakat, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Madrid, Spain